CLINICAL TRIAL: NCT05718999
Title: Development and Internal Validation of a Machine Learning Model to Predict the Occurrence of Incisional Hernia After a Midline Laparotomy
Brief Title: XGBoost for Predict Incisional Hernia
Acronym: XGB&IncHern
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Responsible Party: Principal Investigator, Edgard Lozada, Clinical Research Level D, Hospital Regional de Alta Especialidad del Bajio
Other Study IDs: CI/HRAEB/002/2021; CEI/HRAEB/002/2021 (Other: Hospital Regional of High Speciality of Bajio)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Incisional Hernia: The incisional hernia was defined according to the EHS guidelines as a mass in the abdominal wall with or without a visceral outlet or palpable in the surgical site determined by clinical examination or tomography, this group will present this complication.
  Interventions: Diagnostic Test: Not intervention
- Without Incisional Hernia: The incisional hernia was defined according to the EHS guidelines as a mass in the abdominal wall with or without a visceral outlet or palpable in the surgical site determined by clinical examination or tomography, this group will not present this complication.
  Interventions: Diagnostic Test: Not intervention

INTERVENTIONS:
Diagnostic Test: Not intervention — Not having intervention is an observational study

SUMMARY:
The objective of this study is to develop a predictive model of IH based on machine learning with the use of the XGBoost technique, this will help surgeons in charge of abdominal wall closure to have objective support to determine high-risk patients and in them modify the closure technique or use a mesh according to their choice or the degree of contamination of the abdominal cavity.

DETAILED DESCRIPTION:
Retrospective and observational study. The predictions will make using machine learning models. The programs use the scikit-learn, xgboost and catboost Python packages for modeling.

The evaluation of models will be using fourfold cross-validation, the receiver operating characteristic (ROC) curve, the area under the ROC curve (AUC), and accuracy metrics calculated on the union of the test sets of the cross-validation.

The most critical factors and their contribution to the prediction will identify using a modern tool of explainable artificial intelligence called SHapley Additive exPlanations (SHAP).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Postoperative midline exploratory laparotomy, who underwent urgent or scheduled surgery, regardless of their underlying diagnosis,
* included between January 2010 and December 2016 and who completed 24 months of follow-up after surgery initial surgery.

Exclusion Criteria:

* Reoperated for any cuestion diferent to present of hernia
* Management of open abdomen

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age, postoperative midline exploratory laparotomy, who underwent urgent or scheduled surgery, regardless of their underlying diagnosis, were included between January 2010 and December 2016 and who completed 24 months of follow-up after surgery initial surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Incisional Hernia | 24 months
  incidence of Incisional hernia (the incisional hernia was defined according to the EHS guidelines as: a mass in the abdominal wall with or without visceral outlet or palpable in the surgical site determined by clinical examination or tomography).

SECONDARY OUTCOMES:
Facial dehiscence | 30 days
  Incidence of fascial dehiscence (the fascial dehiscence is the presentation of separation of fascie with leakage of contents from the abdominal cavity

CONTACTS AND LOCATIONS:
Overall Officials: Edgard Efren Lozada Hernández, Principal Investigator — Hospital Regional Of High Speciality of Bajio
Locations (1):
- Hospital regional de Alta Especialidad del bajio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Once the database to be analyzed is identified, the presence of other researchers will be verified to certify the veracity of the data.

REFERENCES:
- [Result] Deerenberg EB, Harlaar JJ, Steyerberg EW, Lont HE, van Doorn HC, Heisterkamp J, Wijnhoven BP, Schouten WR, Cense HA, Stockmann HB, Berends FJ, Dijkhuizen FPH, Dwarkasing RS, Jairam AP, van Ramshorst GH, Kleinrensink GJ, Jeekel J, Lange JF. Small bites versus large bites for closure of abdominal midline incisions (STITCH): a double-blind, multicentre, randomised controlled trial. Lancet. 2015 Sep 26;386(10000):1254-1260. doi: 10.1016/S0140-6736(15)60459-7. Epub 2015 Jul 15. PMID 26188742
- [Result] Jairam AP, Timmermans L, Eker HH, Pierik REGJM, van Klaveren D, Steyerberg EW, Timman R, van der Ham AC, Dawson I, Charbon JA, Schuhmacher C, Mihaljevic A, Izbicki JR, Fikatas P, Knebel P, Fortelny RH, Kleinrensink GJ, Lange JF, Jeekel HJ; PRIMA Trialist Group. Prevention of incisional hernia with prophylactic onlay and sublay mesh reinforcement versus primary suture only in midline laparotomies (PRIMA): 2-year follow-up of a multicentre, double-blind, randomised controlled trial. Lancet. 2017 Aug 5;390(10094):567-576. doi: 10.1016/S0140-6736(17)31332-6. Epub 2017 Jun 20. PMID 28641875
- [Result] Muysoms FE, Antoniou SA, Bury K, Campanelli G, Conze J, Cuccurullo D, de Beaux AC, Deerenberg EB, East B, Fortelny RH, Gillion JF, Henriksen NA, Israelsson L, Jairam A, Janes A, Jeekel J, Lopez-Cano M, Miserez M, Morales-Conde S, Sanders DL, Simons MP, Smietanski M, Venclauskas L, Berrevoet F; European Hernia Society. European Hernia Society guidelines on the closure of abdominal wall incisions. Hernia. 2015 Feb;19(1):1-24. doi: 10.1007/s10029-014-1342-5. Epub 2015 Jan 25. PMID 25618025
- [Result] Deerenberg EB, Henriksen NA, Antoniou GA, Antoniou SA, Bramer WM, Fischer JP, Fortelny RH, Gok H, Harris HW, Hope W, Horne CM, Jensen TK, Kockerling F, Kretschmer A, Lopez-Cano M, Malcher F, Shao JM, Slieker JC, de Smet GHJ, Stabilini C, Torkington J, Muysoms FE. Updated guideline for closure of abdominal wall incisions from the European and American Hernia Societies. Br J Surg. 2022 Nov 22;109(12):1239-1250. doi: 10.1093/bjs/znac302. PMID 36026550
- [Result] Lozada-Hernandez EE, Mayagoitia-Gonzalez JC, Smolinski-Kurek RL, Montiel-Hinojosa L, Hernandez-Villegas L, Morales-Vargas JM, Perez-Sanchez KD, Orozco-Mosqueda A, Cano-Rosas M. Prevention of incisional hernia with a reinforced tension line (RTL) versus primary suture only in midline laparotomies: 3-year follow-up in a randomized clinical trial. Hernia. 2022 Apr;26(2):447-456. doi: 10.1007/s10029-020-02338-9. Epub 2021 Jan 5. PMID 33398464
- [Result] Veljkovic R, Protic M, Gluhovic A, Potic Z, Milosevic Z, Stojadinovic A. Prospective clinical trial of factors predicting the early development of incisional hernia after midline laparotomy. J Am Coll Surg. 2010 Feb;210(2):210-9. doi: 10.1016/j.jamcollsurg.2009.10.013. PMID 20113942
- [Result] Cao GW, Yang WG, Du P. [Observation of the effects of LAK/IL-2 therapy combining with Lycium barbarum polysaccharides in the treatment of 75 cancer patients]. Zhonghua Zhong Liu Za Zhi. 1994 Nov;16(6):428-31. Chinese. PMID 7720497